CLINICAL TRIAL: NCT04799730
Title: Study of CD184 in Systemic Lupus Erythematosus
Brief Title: Expression of CXCR4 in Patients With Systemic Lupus Erythematosus
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Asmaa Abdelfattah Ibrahim, the Master Degree in Clinical and Chemical Pathology, Sohag University
Other Study IDs: Soh-Med-21-03-01
Record Dates: First submitted 2021-03-14; First posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Systemic Lupus Erythematosus
Keywords: CXCR4,CD184,Flow cytometry ,Systemic lupus erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — patient's peripheral-blood mononuclear cells (PBMCs) will be isolated from heparinized venous blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- SLE cases in remission: according to SLE Disease Activity Index (SLEDAI) inactive disease will be considered as SLEDAI <5
- SLE cases in activity: according to SLE Disease Activity Index (SLEDAI) Active disease will be defined as SLEDAI ≥ 5
- Control group: Healthy age and sex matched subjects.

SUMMARY:
The objective of this study is to estimate the possible role of CD184 in the pathogenesis of SLE; comparing its level among SLE cases to healthy controls.

DETAILED DESCRIPTION:
Detection of CXCR4 (CD184) expression on CD19+ B cells by flow cytometry in patients of SLE, comparing its level in the development of lupus activity and pathogenic process of SLE internal organ involvement/ mucocutaneus and/or musculoskeletal involvement. Identify this correlation will be useful for clarifying other accessory factors to improve the diagnosis, better treatment strategy, follow up as well as prognosis for these patients

ELIGIBILITY:
Inclusion Criteria:

* Confirmed SLE patients diagnosed and fulfilled the SLE classification criteria according to the 2019 ACR/EULAR classification criteria for SLE (Aringer et al., 2019)
* Willing and agreed to be included in the study.

Exclusion Criteria:

* Childhood SLE.
* SLE-patients will refuse to consent to this study.
* Other autoimmune diseases.
* Known or suspected malignancies, especially B cell lymphoma.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Study population will be classified into two group:
  1. SLE patients group: Confirmed SLE patients diagnosed and fulfilled the SLE classification criteria according to the 2019 ACR/EULAR classification criteria for SLE (Aringer et al., 2019).
  2. Control group: Healthy age and sex matched subjects.
  Then SLE group I patients will be subdivided according to the disease activity to three subgroups:
  I. Group A: SLE cases in remission II. Group B: SLE cases in activity, but no internal organ involvement (i.e. only mucocutaneus and/or musculoskeletal involvement).
  III. Group C: SLE cases in activity, and with internal organ involvement (renal, neuropsychiatric, hematological or cardiopulmonary).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
changes in the expression of CD184(CXCR4) expression in circulating B cells | 6 months
  Flow cytometry analysis of chemokine receptor (CXCR4):Human peripheral-blood mononuclear cells (PBMCs) labeling with CXCR4 antibody will be performed in the same day after taking blood samples and subsequent measurement of the CXCR4 mean fluorescence intensity (MFI) by flow cytometry. MFI of the anti-chemokine receptor (CXCR4) staining will be calculated according to statistical thresholds set in reference to staining with negative control antibodies. The patient's CXCR4 on CD19+ B cells expression or mean MFI will be further compared to the MFI of the simultaneously performed age-matched controls samples and other subgroups of SLE patients.